CLINICAL TRIAL: NCT02504086
Title: Online Support for Diabetes Self-Management
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Difficulty recruiting participants
Sponsor: University of British Columbia (Other)
Collaborators: University of Minnesota (Other)
Responsible Party: Principal Investigator, Leanne Currie, Associate Professor, University of British Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: F14-01764
Record Dates: First submitted 2015-06-24; First posted 2015-07-21 (Estimated); Last update posted 2016-07-19 (Estimated); Status verified 2016-07

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Online Support (Experimental): 3 months online support, including access to online personal health record and 2.5 hours of online video teleconsultations with certified health professionals
  Interventions: Behavioral: Online Support

INTERVENTIONS:
Behavioral: Online Support — 3 months online support, including access to online personal health record and 2.5 hours of online video teleconsultations with certified health professionals

SUMMARY:
The purpose of this study is to evaluate the effect of online support for diabetes self-management for patients with Type II diabetes in the Vancouver region. Patients will be invited to receive 8 online video consultations (total 2.5 hours) with certified healthcare providers (video calls in a secure Website). Participants will also have access to the use of an online personal health record -- a place to store healthcare information for the patient and healthcare provider to view. Patients' ability to care for their diabetes will be measured at the beginning and the end of the study. Additional measures include glycaemic control, BMI, waist circumference, diabetes self-efficacy, computer and health literacy, patient satisfaction with care and perceived ease of use and perceived usefulness of the technology.

DETAILED DESCRIPTION:
Purpose:

The purpose of this study is to evaluate the effectiveness of a 3-month control-theory-based online support intervention consisting of 8 online video teleconsultations and access to a secure online personal health record on self-management behaviours of adults with type 2 diabetes, as measured by the Summary of Diabetes Self-Care Activities (SDSCA). Secondary outcomes will include glycemic control, BMI, waist circumference, diabetes self-efficacy, computer and health literacy, patient satisfaction with care and perceived ease of use and perceived usefulness of the technology.

Hypothesis:

Patients who receive online support for diabetes self-management and access to an online personal health record will have higher self-management of diabetes scores after they receive the intervention compared to before the intervention.

Justification:

In British Columbia (BC), an estimated 10.3 percent of the population is expected to have diabetes by 2020, at an estimated cost to the BC healthcare system of 1.9 billion dollars per year. Enhancing diabetes self-management has been estimated to be the single most cost-effective intervention in the primary care setting. Results of telemedicine interventions for management of diabetes have been mixed; many interventions show promising improvement in health behaviours, self-efficacy and glycaemic control, while others show small or no effects. A 2015 meta-analysis of the clinical effectiveness of telemedicine randomized controlled trials for type 2 diabetes found a significant decrease in HbA1C overall, with the largest decrease being amongst Internet-based interventions. A recent Cochrane systematic review and meta-analysis of computer-based self-management interventions for adults with type 2 diabetes found that interventions using mobile phones showed a greater reduction in glycaemic control than did the telehealth interventions overall. A meta-regression of techniques in 122 healthy eating and physical activity self-management interventions for diabetes found that self-monitoring explained the greatest amount of among-study heterogeneity, accounting for 13% of these differences. Self-monitoring is a component of control theory, which proposes that in order to effectively manage behaviour, there must be a clear, realistic goal, an action plan for attaining it, a means of monitoring whether a person is on track, feedback, and opportunities for reviewing goals in the light of feedback. Providing additional information for behavioural providers through an online personal health record, and integrating behavioural support with ongoing primary care through shared action plans, the effectiveness of behavioural support provided online may be increased. Standard treatment primarily involves management of diabetes through medications and may involve referral to a diabetes education centre for education about diabetes self-management. The best method to support patient self-management has not been clearly identified.

Objectives:

The specific outcome to be examined is self-management of type II diabetes as measured by the Summary of Diabetes Self-Care Activities (SDSCA).

Research Method:

A pre-post intervention study with a multicentre cohort of 125 patients who will be provided with an online support intervention and followed over three months to evaluate change in diabetes self-management behaviours and clinical outcomes. We will recruit a total of 125 patients with type 2 diabetes through 12 participating primary care physicians. After consent is obtained, participants will be provided with training to use the glucometer, online video teleconsultation tools and online personal health record.

Online Support Intervention:

The online support intervention is designed as a supplement to usual care provided by the family physician, and will be delivered via the Internet through the company Treatment, Inc. a West Vancouver-based provider of patient self-care solutions and services (see Treatment Diabetes Screen shots). The three-month online support intervention involves two primary components to facilitate patient self-management: 8 online video teleconsultations with a certified health professional (for a total of 2.5 hours, weekly at first, then bi-monthly) and access to an online personal health record to promote health care behavioural change. Certified healthcare professionals will provide the 8 online video teleconsultations and will provide reports to the primary care provider as needed and at the end of the 3-month intervention. Participants will also be given a glucose meter (Bayer Contour® Next meter) from which glucose readings can be uploaded to the online personal health record. The patient will use their own glucometer strips as provided by the BC government prescription plan.

Data Collection:

The primary outcome is change in diabetes self-management behaviour as measured by the Summary of Diabetes Self-Care Activities (SDSCA) which includes diet, exercise, self-monitoring of blood glucose, foot care and smoking. Secondary outcomes include change in HbA1C, BMI and waist circumference, diabetes self-efficacy, satisfaction with care, and acceptance of using technology for online support. (See attached document: Measurement Instruments) The primary care provider will have access to the patient's online information, including self-monitored glucose values, for review. Participants will complete online questionnaires at baseline and at end of study.

Sample Size Calculation:

The statistical power for the study was modeled with a two-tailed paired sample t-test to test changes in SDSCA from baseline to three months. Published studies using the SDSCA have shown effects sizes of change in intervention groups ranging from .278 to .53. Thus, conservatively estimating an effect size of .278, to achieve 80% power at a p <.05 significance level, a sample of 125 participants will be required, assuming a 20% longitudinal attrition rate. Attrition rates in the 10% to 20% range have been reported in previous similar Web-based intervention studies.

Data Analysis:

Two-tailed paired sample t-tests will be performed to test for changes in mean self-management behaviours from baseline to three months. Correlations will explore relations between the outcome variables and health literacy, computer literacy and the control variables. Changes across time in the secondary outcomes (clinical outcomes, diabetes self-efficacy) will also be examined using paired-sample t-tests to explore for trends and effect sizes for future studies. All tests will be performed using SPSS version 23, with a p <.05 significance level.

ELIGIBILITY:
Inclusion criteria:

* Men and women 18 years to 80 years
* Current diagnosis of Type 2 Diabetes diagnosed at least 6 months previous to the intervention
* Have seen their participating family physician of the Vancouver Coastal Health Authority catchment area at least twice over the last two years, with at least one of those visits including the code for diabetes.
* English Speaking
* Ability to review the consent form independently
* Have access to the online video teleconsultation and personal health record from their home
* Have basic computer literacy (use a computer and the internet at least once a week)

Exclusion criteria:

* Physical disability that precludes normal internet use
* Diagnosis of a terminal illness
* Pregnancy, planning a pregnancy, or currently lactating

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2015-08; Primary Completion 2016-08 (Estimated); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Change in diabetes self-management behaviours as measured by Summary of Diabetes Self Care Activities (SDSCA; Toobert et al 2000) | baseline and 3 months
  as measured by Summary of Diabetes Self Care Activities (SDSCA; Toobert et al 2000)

SECONDARY OUTCOMES:
Change in glycemic control as measured by HbA1C | baseline and 3 months
  as measured by HbA1C
Change in body mass index as calculated by patient self-reported height and weight | baseline and 3 months
  as calculated by patient self-reported height and weight
Change in waist circumference as measured by patient using provided instructions | baseline and 3 months
  as measured by patient using provided instructions
Change in Diabetes Self-Efficacy as measured by Diabetes Empowerment Scale, short-form (Anderson et al., 2003) | baseline and 3 months
  as measured by Diabetes Empowerment Scale, short-form (Anderson et al., 2003)
Change in Patient Satisfaction with Care as measured by Patient Assessment of Chronic Illness Care (PACIC)(Glasgow et al., 2005; Schmittdiel et al., 2008) | baseline and 3 months
  as measured by Patient Assessment of Chronic Illness Care (PACIC)(Glasgow et al., 2005; Schmittdiel et al., 2008)
Perceived usefulness and perceived ease of use of online support as measured by the Unified Theory of the Acceptance and Use of Technology (UTAUT) for telehealth (Kohnke et al., 2014 based on Venkatesh et al., 2003) | 3 months
  as measured by the Unified Theory of the Acceptance and Use of Technology (UTAUT) for telehealth (Kohnke et al., 2014 based on Venkatesh et al., 2003)

CONTACTS AND LOCATIONS:
Overall Officials: Leanne Currie, PhD, Principal Investigator — University of British Columbia
Locations (1):
- Vancouver primary care offices, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No